CLINICAL TRIAL: NCT03532711
Title: A Study to Characterize and Evaluate Biomarkers of Chemotherapy in Patients With Metastatic Colorectal Cancer In The First-line Setting
Brief Title: Potential Predictive Biomarkers in Patients Undergoing First-line Chemotherapy for Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Wen Zhang, Dr, Fudan University
Other Study IDs: FUSCC-BiomarkerCRC
Record Dates: First submitted 2018-05-04; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Colorectal Cancer; Chemotherapy Effect; Biomarker
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Capecitabine; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chemotherapy: FOLFOX/XELOX/FOLFIRI
  Interventions: Drug: fluorouracil

INTERVENTIONS:
Drug: fluorouracil — chemotherapy treated patients
  Other Names: capecitabine; irinotecan hydrochloride; leucovorin calcium; oxaliplatin; laboratory biomarker analysis

SUMMARY:
Chemoresistance remains an obstacle in treating people with metastatic colorectal cancer (mCRC). Studying samples of blood and tumor tissue in the laboratory from patients with mCRC receiving chemotherapy may help doctors understand the effect of chemotherapy on biomarkers. It may also help doctors predict how patients will respond to treatment. In this study, we aimed to evaluate biomarkers in chemotherapy regimens for first-line chemotherapy for mCRC.

ELIGIBILITY:
Inclusion Criteria Histologically confirmed metastatic colorectal cancer Unresectable metastatic disease must be confirmed histologically if > 2 years since primary diagnosis Measurable metastatic disease > 1 cm by spiral CT scan or > 2 cm by other methods Scheduled to receive first-line chemotherapy for metastatic disease Chemotherapy must include fluorouracil, capecitabine, irinotecan hydrochloride, or oxaliplatin Exclusion Criteria Inadequate or unusable tissue as the only tissue available Brain metastases or meningeal disease Contraindication to chemotherapy Pregnant or nursing Other severe pathology that is likely to worsen during therapy Dementia or severely impaired mental condition Geographical or psychological reasons that would preclude treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed metastatic colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 months
  objective response rate

SECONDARY OUTCOMES:
Overall Survival (OS) | 6 months
  overall survival
Progression Free Survival (PFS) | 6 months
  progression free survival

IPD SHARING:
Plan to Share IPD: No